CLINICAL TRIAL: NCT00958724
Title: A Phase 1 Study Of Neratinib (HKI-272) In Combination With Vinorelbine In Japanese Subjects With Advanced Or Metastatic Solid Tumors
Brief Title: Study Evaluating Neratinib In Combination With Vinorelbine In Subjects With Advanced Or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3144A2-1118 / B1891002
Record Dates: First submitted 2009-08-05; First posted 2009-08-13 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: HKI-272; Vinorelbine; Combination; Solid Tumor; Neratinib; Nerlynx; PB-272
MeSH Terms: interventions — neratinib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neratinib and Vinorelbine (Experimental): Neratinib: 240 mg administered daily by mouth continuously, Vinorelbine: 25 mg/m^2 administered IV on Day 1 and 8 of 21 day cycle
  Interventions: Drug: Neratinib; Drug: Vinorelbine

INTERVENTIONS:
Drug: Neratinib
  Other Names: HKI-272; Nerlynx
Drug: Vinorelbine

SUMMARY:
The purposes of this study are to evaluate the safety and tolerability of neratinib in combination with vinorelbine at the maximum tolerated dose (MTD) determined in a previous study, or to determine a lower MTD of the two drugs, as well as to obtain preliminary information on whether the combination of the two drugs has any effect on solid tumors in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic diagnosis of a solid tumor that is not curable with available therapies for which neratinib plus vinorelbine is a reasonable treatment option.
* At least 1 measurable lesion as defined by Response Evaluation Criteria in Solid Tumors.
* Eastern Cooperative Oncology Group performance status of 0 to 2 (not declining within 2 weeks before signing the informed consent form).
* Recovery from all clinically significant AEs related to prior therapies (excluding alopecia).
* Left ventricular ejection fraction within the study site's limits of normal.
* Screening laboratory values within the following parameters:

  * Absolute neutrophil count: 1.5 × 109/L
  * Platelet count: 100 × 109/L
  * Hemoglobin: 9.0 g/dL
  * Serum creatinine: 1.5 × upper limit of normal
  * Total bilirubin: 1.5 × ULN
  * Aspartate aminotransferase and alanine aminotransferase: 2.5 × ULN (<= 5 × ULN if liver metastases are present).
* For women of childbearing potential, a negative urine or serum pregnancy test result before study entry.
* All female and male subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control for the duration of the study and for 28 days after the last dose of test article. A subject is biologically capable of having children if he or she is using contraceptives or if his or her sexual partner is sterile or using contraceptives.

Exclusion Criteria:

* Prior treatment with anthracyclines with a cumulative dose of doxorubicin of >400 mg/m^2, or of epirubicin >800 mg/m^2, or the equivalent dose for other anthracyclines or derivatives.
* Major surgery, chemotherapy, radical (curative intent) radiotherapy, investigational agents, or other cancer therapy within at least 2 weeks before treatment day 1.
* Bone as the only site of disease.
* Active central nervous system metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth. (Subjects with a history of CNS metastases or cord compression are allowable if they have been definitively treated and are off anticonvulsants and steroids for at least 4 weeks before cycle 1 day 1) .
* QT (QTc) interval > 0.47 s or a known history of QTc prolongation or Torsades de Pointes.
* Presence of clinically significant or uncontrolled cardiac disease, including congestive heart failure (New York Heart Association functional classification of =2), angina requiring treatment, myocardial infarction within the past 12 months, or any clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention.
* Pregnant or breastfeeding women. Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom (eg, Crohn disease, malabsorption, or grade 2 diarrhea of any etiology at baseline).
* Inability or unwillingness to swallow tablets (neratinib).
* Preexisting grade 2 or greater motor or sensory neuropathy.
* Subject known to be human immunodeficiency virus seropositive and/or have acute or chronic hepatitis B infection (hepatitis B surface antigen [HBsAg] positive) or hepatitis C infection (anti-HCV positive).
* History of known hypersensitivity to vinorelbine and any of its components.
* Any other cancer within 5 years prior to screening with the exception of contralateral breast carcinoma, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.
* Clinically significant ongoing or recent infection within 2 weeks before treatment day 1.
* Evidence of significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, make the subject inappropriate for this study. Examples include, but are not limited to, serious active infection (ie, requiring intravenous antibiotic or antiviral agent) or uncontrolled major seizure.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (2):
- Japan (2):
  - Shizuoka Cancer Center, Shizuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Nera 240 + Vino 25: Neratinib 240 mg + Vinorelbine 25 mg/m^2
Period: Overall Study
Arm/Group | Nera 240 + Vino 25
Started | 6
Completed | 0
Not Completed | 6
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 6

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Number of participants experiencing DLT of neratinib in combination with vinorelbine in Japanese patients.
Time Frame: From first dose date to 21st day
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 6
participants | 1

2. Secondary Outcome: Best Overall Response
Description: Best Overall Response in Evaluable Population per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From first dose date to progression or last tumor assessment, up to 40 weeks.
Population: Subjects who met eligibility criteria, received at least 2 weeks of continual daily dosing of neratinib, at least 2 doses of vinorelbine, and underwent at least 1 follow-up tumor assessment at 6 weeks, ie, approximately at cycle 2. In the case of disease progression prior to 6 weeks, a clinical assessment of progressive disease was adequate.
Measure: Count of Participants; unit: Participants
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 6
Participants
  Partial Response | 1
  Stable Disease >= 6 weeks | 5
  Stable Disease >= 24 weeks | 1

3. Secondary Outcome: Duration of Objective Response
Description: The duration of objective response was measured from the time at which measurement criteria were met for Complete Response (CR) or Partial Response (PR) (whichever status was recorded first) until the first date on which recurrence or Progressive Disease (PD) was objectively documented, taking as reference for PD the smallest measurements recorded since the treatment started.
Time Frame: From first response date to PD/death, up to 40 weeks.
Population: Subjects who had a partial or complete response
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 1
weeks | 12.0 [NA to NA] — Confidence Interval not estimable with only 1 subject.

4. Secondary Outcome: Objective Response Rate (ORR)
Description: Proportion of subjects who achieved complete response or partial response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From first dose date to progression or last tumor assessment, up to 40 weeks.
Population: Safety population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 6
percentage of participants | 16.7 [0.4 to 64.1]

5. Secondary Outcome: Progression Free Survival
Description: Number of weeks between the date of the first dose of test article and the first date of disease recurrence or progression, or death due to any cause, was documented, censored at the last evaluation, investigator assessment.
  Disease Progression (PD) is defined using Response Evaluation Criteria in Solid Tumors Criteria (v1.0), at least a 20% increase in the sum of the longest diameters (LD) of target lesions, taking as reference the nadir LD, meaning the smallest sum of the LDs recorded since the treatment started; or unequivocal progression of existing nontarget lesions; or the appearance of any new lesions.
Time Frame: From first dose to last evaluation, up to 40 weeks.
Population: Subjects who met eligibility criteria, received at least 2 weeks of continual daily dosing of neratinib and at least 2 doses of vinorelbine, and underwent at least 1 follow-up tumor assessment at 6 weeks, i.e., approximately at cycle 2. In the case of disease progression prior to 6 weeks, a clinical assessment of PD was adequate.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 6
weeks | 18.2 [18.0 to 24.1]

6. Secondary Outcome: Area Under the Curve (AUC) Tau
Description: AUC of Neratinib at day 8 following administration of Neratinib 240 mg in combination with Vinorelbine 25 mg/m^2 to Japanese Subjects with Cancer.
Time Frame: Predose, and hour 1, 2, 4, 6, 8 and 24 on day 8.
Population: Population for pharmacokinetic analyses consisted of all subjects in this study who received at least 1 dose of neratinib and provided samples for pharmacokinetic assessments.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 5
ng*hr/mL | 1330 (925)

7. Secondary Outcome: Terminal-phase Elimination Half-life
Description: Terminal-phase elimination half-life of Neratinib at day 8 following Administration of Neratinib 240 mg in combination with Vinorelbine 25 mg/m^2 to Japanese Subjects with Cancer.
Time Frame: Predose, and hour 1, 2, 4, 6, 8 and 24 on day 8.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Nera 240 + Vino 25
Number analyzed (Participants) | 4
hr | 14.37 (3.41)

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to 40 weeks.
Arm/Group | Nera 240 + Vino 25
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nera 240 + Vino 25 (N=6)
Peritoneal abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nera 240 + Vino 25 (N=6)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 6
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 6
Left ventricular dysfunction (Cardiac disorders) | 1
Keratitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Face oedema (General disorders) | 1
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 2
Proctitis infectious (Infections and infestations) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood chloride decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Monocyte count decreased (Investigations) | 1
Protein urine (Investigations) | 1
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Vasculitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less